CLINICAL TRIAL: NCT06074484
Title: An Open-label, Single-arm, Multi-center, Phase II Study to Evaluate the Efficacy and Safety of RC48-ADC Combined With AK104 in Perioperative Treatment of Muscle-Invasive Bladder Cancer
Brief Title: A Study of RC48-ADC Combined With AK104 For Perioperative Treatment of Muscle-Invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Shanxi Province Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCVDUCIIR012
Record Dates: First submitted 2023-08-22; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-08

CONDITIONS: Muscle Invasive Bladder Carcinoma
Keywords: RC48-ADC; AK104
MeSH Terms: interventions — disitamab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC +AK104 (Experimental): Participants received 4 preoperative cycles of RC48-ADC（2.0 mg/kg，Q2W） plus AK104（6.0 mg/kg，Q2W）, followed by surgery, followed by up to 14 cycles of postoperative AK104（10 mg/kg，Q3W）and 6 cycles of postoperative RC48-ADC（2 mg/kg，Q3W）
  Interventions: Drug: RC48-ADC; Drug: AK104

INTERVENTIONS:
Drug: RC48-ADC — 4 preoperative cycles of RC48-ADC （2.0 mg/kg，intravenous (IV) infusion，Q2W）, followed by surgery, followed by up to 6 cycles of postoperative RC48-ADC（2.0 mg/kg，intravenous (IV) infusion，Q3W）
  Other Names: Disitamab Vedotin
Drug: AK104 — 4 preoperative cycles of AK104（6.0 mg/kg，intravenous (IV) infusion，Q2W）, followed by surgery, followed by up to 14 cycles of postoperative AK104（10 mg/kg，intravenous (IV) infusion，Q3W）
  Other Names: Cadonilimab Injection

SUMMARY:
This study will evaluate the efficacy and safety of intravenous RC48-ADC combined with AK104 in perioperative treatment of muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
36 patients with Muscle-invasive Bladder Cancer（MIBC） scheduled for radical cystectomy will participate in this study. The patient had not previously received any antitumor system therapy for MIBC. HER2 expression in MIBC patients is defined as the expression of HER2 in tumor tissues detected by immunohistochemistry (IHC) as IHC 1+, 2+, or 3+. After enrollment, the subjects will receive 4 cycles neoadjuvant therapy and 14 cycles adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years.
* Predicted survival ≥ 12 weeks.
* Histologically confirmed diagnosis of muscle invasive bladder cancer (MIBC) .Naive of antitumor systematic treatment or radiotherapy.
* Have clinically non-metastatic bladder cancer (cT2-T4a, N0-1, M0) determined by imaging. Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years.
* Predicted survival ≥ 12 weeks.
* Histologically confirmed diagnosis of muscle invasive bladder cancer (MIBC).Naive of antitumor systematic treatment or radiotherapy.
* Have clinically non-metastatic bladder cancer (cT2-T4a, N0-1, M0) determined by imaging.
* Be deemed eligible for Radical Cystectomy (RC) + Pelvic Lymph Node Dissection (PLND).
* HER2 expressing (i.e. IHC 1+ 2+ or 3+) as confirmed by the local lab.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function, evidenced by the following laboratory results within 7 days prior to the study treatment.
* Male and female participants are eligible to participate if they agree to the contraception use as per study protocol.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.
* Be deemed eligible for Radical Cystectomy (RC) + Pelvic Lymph Node Dissection (PLND).
* HER2 expressing (i.e. IHC 1+ 2+ or 3+) as confirmed by the local lab.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function, evidenced by the following laboratory results within 7 days prior to the study treatment.
* Male and female participants are eligible to participate if they agree to the contraception use as per study protocol.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Has received other antitumor therapy before planned start of trial treatment.
* History of major surgery within 4 weeks of planned start of trial treatment.
* Diagnosed with HBsAg, HBcAb positive and HBV DNA copy positive, or HCVAb positive, or HIVAb positive.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* NYHA Class III heart failure.
* Suffering from active infection requiring systemic treatment.
* Uncontrolled hypertension, diabetes, Interstitial lung Disease, or COPD;
* Treated with systemic treatment (e.g. immunomodulators, corticosteroids or immunosuppressants) for the autoimmune disease within 2 years prior to the study treatment.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Pregnancy or lactation.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-08-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | Up to approximately 16 Weeks (Time of surgery)
  pCR rate is defined as the percentage of participants having pCR. pCR is defined as absence of viable tumor (pT0pT0N0) in examined tissue from RC and PLND.

SECONDARY OUTCOMES:
Rate of Pathologic Response | Up to approximately 16 Weeks (Time of surgery)
  No residual tumor (ypT0N0) and partial response (ypTis-1N0) in surgical specimen.
1-3 year Disease Free Survival Rate | From approximately 12 Months up to approximately 36 Months
  The percentage of participants disease free on 1-3 year after surgery.
Objective Response Rate (ORR) | Up to approximately 16 Weeks
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Overall Survival (OS) | Up to approximately 60 Months
  Overall survival is defined as the time from enrollment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Nianzeng Xing, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China